CLINICAL TRIAL: NCT04651192
Title: Neurological and Psychological Effects of Combat-Related Stress
Status: Completed | Type: Observational
Sponsor: Tel Aviv University (Other)
Collaborators: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Other Study IDs: TAUatm
Record Dates: First submitted 2020-11-24; First posted 2020-12-03 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Stress Disorder, Posttraumatic; Stress, Psychological
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress, Psychological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Soldiers: 50 Israeli Defense Forces (IDF) infantry soldiers, all male, aged 18 years, with Hebrew as the dominant language and no condition excluding an MRI scan.
  Interventions: Other: Combat Exposure
- Students: 50 Reserve Officer Training Corps (ROTC) undergraduate students at Tel-Aviv University, all male, aged 18-19, with Hebrew as the dominant language and no condition excluding an MRI scan.

INTERVENTIONS:
Other: Combat Exposure — Soldiers will be exposed to combat as part of their routine military service. The ROTC students will not be exposed to combat.
  Groups: Soldiers

SUMMARY:
The purpose of this study is to determine what is the neurological and cognitive impact of combat exposure and prolonged stress, in the form of service in the Israeli Defense Forces.

DETAILED DESCRIPTION:
Attention biases in threat processing have been assigned a prominent role in the etiology and maintenance of anxiety disorders. This study aimed to characterize the mental resilience of combat soldiers, and explore the neuro-cognitive impact of prolonged stress, using eye-tracking, MRI and fMRI measurements. Participants will be assessed using questionnaires, cognitive tasks and magnetic imaging at 5 timepoints over the span of 4 years. Outcome measures will be depression, anxiety and post-traumatic scores, as well as dwell time on threat in eye-tracking paradigms tested in previous studies, and blood oxygen level-dependent (BOLD) signals in magnetic resonance imaging (MRI) measurements.

ELIGIBILITY:
Inclusion Criteria:

* Soldiers in the paratroopers brigade or students in Tel-Aviv University;
* A signed consent form;
* Hebrew native speakers.

Exclusion Criteria:

* A diagnosis of a neurological disorder (i.e., epilepsy, brain injury);
* Drug or alcohol abuse;
* Cannot undergo an MRI scan, due to metal implants or other metallic foreign bodies, claustrophobia, large tattoos or irremovable piercings;
* Require glasses with a number greater than 7;
* A diagnosis of psychotic or bipolar disorders.

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy 18-year-old Israeli males.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline - PTSD Checklist for DSM-5 (PCL-5) score | 4 years, from time point 1 to time point 5
  PCL is questionnaire assessing posttraumatic stress disorder symptoms. It contains 20 items on a severity scale of 0-4, measuring the existence and severity of post-traumatic symptoms. The minimal score, indicating no post-traumatic stress, is 0. The maximal score is 80, indicating extremely severe post-traumatic stress.
Neurological measures - Gray matter volume | 4 years, from time point 1 to time point 5
  Gray matter volume, i.e. the density of brain cells in a particular region (outcome to be measured in cm3), to be derived from the MRI scans, and compared between the two groups across the various time points.
Neurological measures - Functional connectivity | 4 years, from time point 1 to time point 5
  Functional connectivity, indicating the level of synchronous activity of certain brain regions during rest (temporal correlation is usually expressed as a Pearson's r); Also to be derived from the MRI scans, and compared between the two groups across the various time points.
Neurological measures - Structural connectivity | 4 years, from time point 1 to time point 5
  Structural connectivity between regions of the brain (Diffusivity is measured as 10-3mm2.s-1) and the properties of the white matter (expressed with Diffusion tensor imaging (DTI) measures, mainly Fractional Anisotropy (FA) and Mean Diffusivity (MD)); Also be derived from the MRI scans, and compared between the two groups across the various time points.
Neurological measures - Task activations | 4 years, from time point 1 to time point 5
  Task activations, and specifically the areas activated during the dot-probe task, and how they change over time (expressed as the level of the BOLD signal strength change during the task). To be derived from the MRI scans, and compared between the two groups across the various time points.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No